CLINICAL TRIAL: NCT05863247
Title: Ocular Biomarkers for Successful Premium Trifocal Intra-ocular Lenses Implantation
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Hospital dos Lusíadas (Other)
Responsible Party: Principal Investigator, Guilherme Neri Pires, Principal Investigator, Hospital dos Lusíadas
Other Study IDs: HdosLusiadas
Record Dates: First submitted 2023-05-09; First posted 2023-05-17 (Actual); Last update posted 2023-05-19 (Actual); Status verified 2023-05

CONDITIONS: Presbyopia; Low Vision
Keywords: cataract; multifocal IOL
MeSH Terms: conditions — Presbyopia; Vision, Low; Cataract | interventions — Patient Reported Outcome Measures

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- pseudophakic patients with post-operative dysphotpsias: Patients who report dyshoptsias after bilateral in-the-bag implantation of a trifocal intra-ocular lens (AT LISA 839mp)
  Interventions: Other: Patient Reported Outcomes / Biometric data revision
- pseudophakic patients without post-operative dysphotpsias: Patients who don't report dyshoptsias after bilateral in-the-bag implantation of a trifocal intra-ocular lens (AT LISA 839mp)
  Interventions: Other: Patient Reported Outcomes / Biometric data revision

INTERVENTIONS:
Other: Patient Reported Outcomes / Biometric data revision — Multivariate statistical analysis will be done to identify the reported biomarkers to characterize patients into the following categories: satisfied without dysphotopsias, unsatisfied with dysphotopsias, satisfied with dysphotopsias, unsatisfied without dysphotopsias.Main outcome measures will be photic phenomena at 6 months of follow-up in correlation with the following pre-surgical parameters: macular ganglion cell complex thickness and/or total ocular and corneal higher-order aberrations (coma, trefoil, spherical aberration). Patients with known contributing factors for the development of dysphotopsias (such as residual refractive error, IOL decentration, posterior capsular opacification) will be excluded from the analyzis.
  Other Names: AT LISA tri 839MP (Carl Zeiss Meditec AG)

SUMMARY:
The purpose of this study is to identify ocular biomarkers that can predict the success of phacoemulsification with bilateral AT LISA try 839MP (Carl Zeiss Meditec AG) implantation to achieve satisfactory post-post-operativly spectacle-free vision. Social, biometric and patient reported outcomes will be evaluated.

DETAILED DESCRIPTION:
Pre-operatively all patients were submitted to a comprehensive ophthalmic history and examination including, corneal topography, and aberrometry (Pentacam), biometry (IOLMaster 700, Carl Zeiss Meditec AG, Jena, Germany), specular microscopy (CEM 539, Nidek Co Ltd.), and macular and papillary Optical Coherence Tomography (Cirrus 4000 Hd OCT, Carl Zeiss Meditec AG).

All surgeries were performed by the same surgeon done by standard phacoemulsification with in-the-bag IOL placement. Patients had both eyes operated within a week.

Patients were assessed at day 1, 6, and month 3 after surgery. Six months post-operatively, refraction and slit-lamp examination was performed, and patients asked to complete the patient reported outcome questionnaire that evaluates visual satisfaction, spectacle independence and dysphoptsia like-symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 45 years old with clinical identified bilateral cataracts
* Patients that want to have good vision most of the time without glasses at all distances
* Highest limit of mesopic pupil of 6 mm
* Corneal total higher-order aberration (HOA) ≤ 0.5 μm
* Angle kappa ≤ 0.58 mm
* Absence of cornea ectasia diagnostic criteria.

Exclusion Criteria:

* Patients with moderate or severe dry eye syndrome
* Ocular comorbidities such as corneal, retinal or optic nerve disease
* Previous ocular surgeries
* Patients with unreal post-surgical visual expectations
* Patients with known mild cognitive impairment or dementia.

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Included patients presented with bilateral/unilateral cataract and pretended spectacle-free vision for all distances (far , intermediate and near).
Sampling Method: Probability Sample
Enrollment: 154 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Correlation between macular ganglion cell thickness and contrast sensitivity in refractive cataract surgery patients - Identifying cutoff values that predict favourable mIOL adaptation | December 2023
  Evaluate if there is a correlation between macular ganglionar cell complex thickness and post-operative contrast-sensitivity at 6 months post-op
HOA detailed profile impact in dysphotopsia incidence after refractive cataract surgery - - Identifying cutoff values that predict favourable mIOL adaptation | December 2023
  Evaluate if specific HOA have a greater impact and association with dysphotopsias under the same IOL platform at 6 months post-op

CONTACTS AND LOCATIONS:
Overall Officials: Guilherme Pires, MD, Principal Investigator — Hospital dos Lusíadas
Locations (1):
- Hospital dos Lusíadas, Lisbon, Portugal

IPD SHARING:
Plan to Share IPD: No